CLINICAL TRIAL: NCT06994169
Title: Glofitamab in Real Life
Status: Recruiting | Type: Observational
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Other Study IDs: GloRel
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Large B-cell Lymphoma
Keywords: CAR-T; Glofitamab
MeSH Terms: interventions — glofitamab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated in EPA: Patients treated in Expanded Access Program to Glofitamab
  Interventions: Drug: Glofitamab

INTERVENTIONS:
Drug: Glofitamab — Glofitamab received for DLBCL in Early Phase Access

SUMMARY:
To date, more than 300 patients have been treated with Glofitamab in the Expanded Access Programme (EAP) in France. In this study, it is proposed to perform a retrospective analysis of some of these patients. The aim is to describe the efficacy and safety of Glofitamab in the largest reported real-world cohort, with an expected median follow-up of more than 9 months. Particular focus will be given to the relapsed or refractory chimeric antigen receptors-T (CAR-T) population to confirm the response rates (CRR: 35-39%) of Glofitamab in this population and to assess the optimal timing of therapy initiation [8, 15].

ELIGIBILITY:
Inclusion Criteria:

* patient enrolled in the French Glofitamab EAP for R/R DLBCL before 2024 November 1st, 2024
* patient who received at least Obinutuzumab pretreatment and one infusion of Glofitamab
* adult patient
* patient who is informed of the study and who did not oppose to their data collection

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: French patients enrolled in the EAP before 1st of November 2024 and treated with at least Obinutuzumab pretreatment and one infusion of Glofitamab for R/R DLBCL We expect to collect data from 200-250 patients from this population with a minimum of 6 months of follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Best Complete Response Rate (best CRR) during treatment, assessed by investigator according to Lugano 2014 criteria. | 6 months

SECONDARY OUTCOMES:
Complete metabolic response rate and overall response rate (ORR) by investigator assessment according to Lugano 2014 criteria | 1 month, 2 months, 3 months, 6 months
Progression-free survival (PFS) | 6 months
Event-Free Survival (EFS) | 6 months
Overall survival (OS) | 6 months
immune effector cell-associated neurotoxicity syndrome (ICANS) rate | 6 months
≥ grade 2 Cytokine release syndrome (CRS) rate | 6 months
intensive care unit (ICU) admission rate | 6 months
rate and cause of rehospitalization due to an adverse event potentially related to Glofitamab, | 6 months
number of significant medical events leading to hospitalization | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume MANSON, MD, Study Chair — Lymphoma Study Association; Gilles CROCHET, MD, Study Chair — The Lymphoma Academic Research Organisation
Locations (30):
- France (30):
  - CH Victor Dupouy, Argenteuil
  - CH d'Avignon - Hôpital Henri Dufaut, Avignon
  - CH de la Côte Basque, Bayonne
  - CHRU Besançon - Hôpital Minjoz, Besançon
  - Hopital D'Instruction Des Armees Percy, Clamart
  - Hopital Henri Mondor, Créteil
  - CHU de Dijon - Hôpital le Bocage, Dijon
  - CH de Dunkerque, Dunkirk
  - CHU de Grenoble - Hôpital Albert Michallon, La Tronche
  - Hôpital de Libourne, Libourne
  - CHRU de LILLE - Claude Huriez, Lille
  - Hopital Saint Vincent-de-Paul, Lille
  - Centre Léon Bérard, Lyon
  - INSTITUT PAOLI CALMETTES - Service Hématologie, Marseille
  - Clinique du Pont de Chaume, Montauban
  - CH de Mulhouse Sud Alsace, Mulhouse
  - CHR d'Orléans, Orléans
  - Hopital Saint-Louis, Paris
  - Chu de Bordeaux - Hopital Haut-Leveque, Pessac
  - CHU Lyon Sud, Pierre-Bénite
  - CHU de Poitiers - Hôpital de La Milétrie, Poitiers
  - CH de Quimper Cornouaille, Quimper
  - CHU de Rennes - Hôpital de Pontchaillou, Rennes
  - Institut Curie - Site Saint-Cloud, Saint-Cloud
  - CHU de Strasbourg, Strasbourg
  - Institut Universitaire du Cancer de Toulouse - Oncopole, Toulouse
  - Chu Bretonneau, Tours
  - CHRU de Nancy - Hôpital de Brabois, Vandœuvre-lès-Nancy
  - Ch de Bretagne Atlantique, Vannes
  - Gustave Roussy Cancer Campus Grand Paris, Villejuif

IPD SHARING:
Plan to Share IPD: No